CLINICAL TRIAL: NCT07330791
Title: Right Phrenic Nerve Localization Using CT Scanning: Implications for Radiofrequency Ablation Procedures
Brief Title: Right Phrenic Nerve Localization on CT for Ablation
Status: Completed | Type: Observational
Sponsor: Centro Medico Teknon (Other)
Responsible Party: Principal Investigator, Antonio Berruezo, MD, PhD, Chief of Electrophysiology Unit, Centro Medico Teknon
Other Study IDs: Phrenic nerve CT-Localization
Record Dates: First submitted 2025-12-10; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-09

CONDITIONS: We Evaluated CT-guided Localization of the Right Phrenic Nerve to Enhance Safety in Transcatheter Ablation
Keywords: Right Phrenic Nerve; Phrenic Nerve Localization; Computed Tomography; CT-Guided Imaging; Radiofrequency Ablation; Catheter Ablation; Transcatheter Ablation Safety; Cardiac Ablation Complications; Ablation Procedures; Phrenic Nerve Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- This study will enroll patients undergoing two distinct types of ablative procedures g: A total of 80 consecutive patients will be included:
  * 60 patients will be enrolled using a single electric stimulation output set at 20 mA, 2 ms amplitude width and 1000 ms cycle length
  * 20 patients will be enrolled using a double electric stimulation output set respectively at 10 mA and 20 mA (2 ms amplitude width and 1000 ms cycle length)

SUMMARY:
The anatomical location of the right phrenic nerve (RPN) in close proximity to the right pulmonary veins has become a critical consideration for electrophysiologists performing pulmonary vein isolation, the cornerstone treatment for atrial fibrillation. Although radiofrequency ablation in this region is rarely associated with complications-unlike cryoballoon ablation-the proximity of the RPN to the ablation site is considered the most widely accepted mechanism of nerve injury. Therefore, accurately defining its anatomical course is essential to prevent complications.

This concern extends to any ablation procedure performed near the RPN, including those targeting the lateral-posterior region of the right atrium, particularly during atrial tachycardia ablation or cardioneuroablation. Several methods have been used to precisely localize the RPN. The most commonly employed technique is phrenic nerve stimulation; however, there is growing interest in the use of computed tomography (CT) to identify structures running parallel to the nerve-such as the pericardiophrenic artery and vein-enhanced with contrast. Three-dimensional reconstruction through image segmentation has proven useful in defining the anatomy of cardiac chambers and adjacent extracardiac structures.

This study aims to compare two approaches for visualizing the course of the right phrenic nerve: one based on computed tomography imaging and the other on the nerve's response to stimulation during the procedure. This comparison will allow us to assess the concordance between imaging findings and intra-procedural observations, ultimately contributing to improved procedural safety.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Patients who have undergone or will undergo transcatheter AF ablation or CNA
* Availability of 64-slice contrast-enhanced MDCT with RPN segmentation using ADAS® software prior to ablation
* Age ≥ 18 years

Exclusion Criteria:

* Inability to provide informed consent
* Inability to perform contrast-enhanced CT before transcatheter AF ablation or CNA
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients underwent an electrocardiography-gated cardiovascular CT using a 64-slice multidetector row CT scanner (Revolution CT, GE Healthcare Global Diagnostic Imaging) prior to the ablation procedure. The position line was set at 0.5 cm below the tracheal bifurcation to the cardiac diaphragmatic surface. The acquisition was performed within a single breath- hold. The gantry rotation time was 0.35 s, and the tube current was 350-750 mA at 120 kV. Iodinated contrast material (60 mL; Omnipaque 300 mg/mL), was injected at a rate of 4-5 mL/s, followed by 20 mL of saline solution. A second acquisition immediately after is performed to study the venous phase. Original images at 75% or 45% R-R intervals were transferred to post-processing Workstation, with a section thickness of 0.625 mm. If motion artifacts appeared, the electrocardiographic editing technique was used and the reconstructed window was moved forward or backward for 5% R-R interval until the motion artifacts disappeared.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
analyse the anatomy of the RPN | From January 2021 to April 2025
  The primary endpoint of this study is to analyse the anatomy of the RPN using three-dimensional (3D) imaging and iso-distance mapping with ADAS® software, and to validate its accuracy through traditional pace mapping.
Accuracy of Imaging-Guided Anatomical Localization of the Phrenic Nerve with ADAS® software Compared With Conventional Pacemapping | from the procedure to 12 months later
  The positions as observed by the 2 different methods are compared and the correlation was expressed as a percentage. Global image correlation is computed as the mean correlation between methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Antonio Berruezo, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided